CLINICAL TRIAL: NCT05393154
Title: Pilot Study of Biopsy Scanner for Evaluation of Bronchoscopic Small Biopsy Specimens
Brief Title: Pilot Study of Biopsy Scanner for Evaluation of Bronchoscopic Small Biopsy Specimens to Determine Adequacy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aquyre Bioscience, Inc (Industry)
Collaborators: Johnson & Johnson (Industry); Boston University (Other); Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: HEATMAP Lung Biopsy Study
Record Dates: First submitted 2022-05-03; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer
Keywords: Lung Biopsy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Participant: Non-destructive imaging of biopsies using the Aquyre system
  Interventions: Device: Biopsy Adequacy Evaluation by Aquyre Biopsy Scanner

INTERVENTIONS:
Device: Biopsy Adequacy Evaluation by Aquyre Biopsy Scanner — Microscopic viewing and imaging of Bronchoscopic Biopsy Specimens using Full Field Optical Coherence Tomography and Dynamic Cell Imaging

SUMMARY:
The aim of the study is to assess the performance of Aquyre Biopsy Scanner technology (the FDA class I medical device) at determining if tissue from the lymph nodes and lung nodules, taken during a bronchoscopy procedure, is adequate for a diagnosis. The study will assess how well the Aquyre Biopsy Scanner can differentiate between tissue samples that meet certain requirements that allow for further diagnostic analysis and samples that do not.

DETAILED DESCRIPTION:
In this study, lymph node or lung nodule tissue will be collected by bronchoscopy as part of standard clinical care. The tissue is being collected to help make a diagnosis of a pulmonary condition. The same amount of tissue that is collected per standard of care for diagnosis will be collected during the study; no additional tissue is taken for this study. The biopsy sample will be analyzed by the Aquyre Biopsy Scanner which will provide images of unprocessed lung biopsy tissue taken during your procedure. A pathologist will also analyze the tissue sample in accordance with existing clinical guidelines. The doctor will use the pathology results to help make a diagnosis of your condition. The results of the Aquyre Biopsy Scanner analysis will be compared to the pathology results. This will help determine how well the Aquyre Biopsy Scanner performs in identifying tissue samples that are suitable for pathology analysis and those that are not. The comparison between Aquyre Biopsy Scanner and the pathology analysis is the experimental part of the study.

The tissue will not be collected specifically for study purposes. Rather, the tissue will be collected as part of the existing clinical care. The same amount of tissue that is collected per standard of care for diagnosis will be collected during the study, the study does not require additional tissue. In addition, the biopsy samples will be divided so the evaluation of the tissue by the pathologist will also be performed, which is part of standard clinical care.

The Aquyre microscope is non-destructive, therefore the tissue samples will be available for subsequent pathology analysis using standard techniques. The experimental part of this study is to compare the images from the microscope to the reading/diagnosis from the pathologist.

NOTE: According to NIH definition, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4083571/ this is an observational study design, which evaluate the accuracy of diagnostic procedures and tests as compared to other diagnostic measures. Diagnostic results of the Aquyre microscope are used for observational comparison only, and not used to direct or change patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study procedures.
2. Patient has a radiographically identified lung lesion(s) suspicious for malignancy and requiring histopathologic diagnosis.
3. Patient with a previously obtained (within 3 months) CT image showing at least one solid lesion equal to or greater than 1 cm in diameter or at least one semisolid lesion with a solid component of equal to or greater than 1 cm in diameter.
4. Bronchoscopic biopsy procedure is planned for the above lesion(s).

Exclusion Criteria:

1. Patient does not meet the requirements to undergo biopsy as determined by the treating physician.
2. Patient is unable to provide a signed informed consent to participate in the study.
3. Patient has only ground glass lesion(s) that do not have a solid component.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tissue will be collected from patients with radiographically identified lung lesions suspicious for cancer for whom a biopsy is being performed for pathological diagnosis, as determined by the investigator.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The performance characteristics (sensitivity, specificity, PPV, and NPV) will be calculated for the Aquyre Biopsy Scanner image relative to Pathology. | through study completion, an average of 1 year
  Evaluation of Aquyre Biopsy images by the bronchoscopist to determine biopsy adequacy comparing to results of pathology.

SECONDARY OUTCOMES:
Test characteristics will be calculated for the ROSE slides relative to Pathology. | through study completion, an average of 1 year
  Evaluation of Aquyre Biopsy images by the bronchoscopist to determine biopsy adequacy comparing to results of ROSE slides

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Billatos, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States